CLINICAL TRIAL: NCT07156604
Title: Vebreltinib for Neoadjuvant Treatment in Patients With Stage IIA-IIIB (N2) Non-small Cell Lung Cancer (NSCLC) Harboring METex 14 Skipping Mutant
Brief Title: Vebreltinib for Neoadjuvant in METex 14 Skipping Mutant Stage IIA-IIIB (N2) Non-small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Chief of Thoracic Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP--1033
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: NSCLC; Neoadjuvant Therapy
Keywords: Vebreltinib; METex 14 skipping mutant; neoadjuvant treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vebreltinib Arm (Experimental): treated with Vebreltinib (200 mg bid po) for 8 weeks before surgery. The subjects were evaluated by the investigators and the surgical resection was performed within approximately 2 weeks after the neoadjuvant treatment.
  Interventions: Drug: Vebreltinib Enteric Capsules

INTERVENTIONS:
Drug: Vebreltinib Enteric Capsules — treated with Vebreltinib (200 mg bid po) for 8 weeks before surgery.

SUMMARY:
This is a prospective, single-center phase II clinical study aimed at evaluating the efficacy and safety of Vebreltinib in neoadjuvant treatment for patients with resectable stage IIA-IIIB (N2) non-small cell lung cancer (NSCLC) with MET exon 14 skipping mutations. In the study, all eligible subjects who signed the informed consent and met the inclusion and exclusion criteria were treated with Vebreltinib (200 mg bid po) for 8 weeks before surgery. The subjects were evaluated by the investigators and the surgical resection was performed within approximately 2 weeks after the neoadjuvant treatment. The study used RECIST v1.1 for imaging assessment. A CT or enhanced CT scan was conducted within 2 weeks after the end of treatment, and then every 180 days (±14) after surgery until 3 years, and then annually until disease recurrence or death, or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient shall sign the Informed Consent Form.
* Aged 18 ≥ years.
* Histological or cytological diagnosis of NSCLC by needle biopsy, and evaluated by researchers as stage IIA-IIIB(N2).
* NGS gene testing confirmed MET exon 14 skipping mutations (NGS results from tissue or blood samples certified by CLIA or CAP-approved laboratories);
* Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
* According to the MDT evaluation (which should include a thoracic surgeon specializing in tumor surgery), it is considered that the primary NSCLC is potentially completely resectable;
* At least 1 measurable lesion according to RECIST 1.1.
* Patients with good function of other main organs (liver, kidney, blood system, etc.)
* Patients with lung function can tolerate surgery;
* Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
* Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 d

Exclusion Criteria:

* Previously received targeted therapy (including TKI or monoclonal antibodies), immunotherapy, or any investigational drug treatment for NSCLC;
* Pathological confirmation of mixed small cell and non-small cell lung cancer;
* Patients with a malignancy other than NSCLC within five years prior to the start of this trial，except for cured basal cell carcinoma of the skin, early gastrointestinal (GI) carcinoma excised through endoscopy, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, or any cured cancer deemed to have no impact on the survival of the current NSCLC;
* Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;
* Patients with congenital or acquired immune dysfunction (such as HIV infected individuals);
* Received other major surgical treatments (excluding diagnosis) within 4 weeks prior to the start of the study or expected to undergo major surgical treatments during the study period;
* Participants who are allergic to the test drug or any auxiliary materials; 8.A history of extensive diffuse bilateral interstitial fibrosis in the past or before medication, or a known grade 3 or 4 history of interstitial fibrosis or interstitial lung disease, including pneumonia, allergic pneumonia, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not including local radiation pneumonia or radiation pulmonary fibrosis history;
* Pregnant or lactating women;
* Any malabsorption;
* Participants suffering from nervous system diseases or mental diseases that cannot cooperate
* Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) rate | Up to 30 months
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants.

SECONDARY OUTCOMES:
Objective response (ORR) rate | up to 30 months
  orr is defined as the proportion of patients who achieve partial response (PR), or complete response (CR) among all patients.
Disease control rate (DCR) | up to 30 months
  DCR Rate is defined as the proportion of patients who achieve stable disease (SD), partial response (PR), or complete response (CR) among all patients.
Pathologic complete response (PCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.
Event-free survival (EFS) | up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
3-year overall survival Rate | Up to 36 months
  OS is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Overall survival (OS) | up to 60 months
  OS is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan CHEN, phd, Principal Investigator — Fudan University Shanghai Cancer Center, Shanghai,
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai,, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided